CLINICAL TRIAL: NCT05985850
Title: Evaluating Tetrahydrocannabinol as an Adjunct to Opioid Agonist Therapy for Individuals Living With Opioid Use Disorder: A Phase II, Placebo-controlled, Blinded, Pilot Study to Assess Safety and Feasibility (THC-MMT)
Brief Title: Evaluating Tetrahydrocannabinol as an Adjunct to Opioid Agonist Therapy
Acronym: THC-MMT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BC Centre on Substance Use (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, M. Eugenia Socias, Assistant Professor, Department of Medicine, UBC; Research Scientist, BCCSU, BC Centre on Substance Use
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCCSU-005
Record Dates: First submitted 2023-07-26; First posted 2023-08-14 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Opioid Use Disorder; Methadone; Cannabis; Fentanyl
Keywords: addiction; Opioid Use Disorder; Cannabis; Harm Reduction; Opioid; Pain; Quality of Life; Cannabidiol
MeSH Terms: conditions — Opioid-Related Disorders; Marijuana Abuse; Behavior, Addictive; Harm Reduction; Pain

STUDY DESIGN:
Intervention Model Description: Phase 1: 1:1 randomization Phase 2: Open-label
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aurora 1:1 Drops (Indica) (Experimental): Aurora 1:1 Drops (Indica)
  Balanced 1:1 ratio of THC and CBD packaged in a 30 mL bottle:
  THC: 16.8 mg/g (+/- 15%) CBD: 16.8 mg/g (+/- 15%)
  Induction and dosing will be ad libitum and sublingually self-administered. Initial dose will be 5 mg (equivalent to 0.25 mL)/day and participants will be able to titrate in increments of 2.5mg (0.125 mL)/day up to a maximum of 40 mg (2 mL)/day, in consultation with a study physician.
  Interventions: Drug: Aurora 1:1 Drops (Indica)
- Placebo (Placebo Comparator): Formulated using the same medium chain triglyceride (MCT) oil as Aurora 1:1 Drops (Indica)
  Induction and dosing will be ad libitum and sublingually self-administered. Initial dose will be 5 mg (equivalent to 0.25 mL)/day and participants will be able to titrate in increments of 2.5mg (0.125 mL)/day up to a maximum of 40 mg (2 mL)/day, in consultation with a study physician.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aurora 1:1 Drops (Indica) — Aurora 1:1 Drops (Indica) is created by extracting cannabinoids and terpenes and the concentrated extract is then diluted in medium-chain triglyceride (MCT) oil for optimal use.
  Arms: Aurora 1:1 Drops (Indica)
Drug: Placebo — Medium-chain triglyceride (MCT) oil with the same appearance, color, and taste as the Aurora 1:1 Drops (Indica).
  Arms: Placebo

SUMMARY:
This pilot study will evaluate the feasibility and safety of using 1:1 tetrahydrocannabinol (THC):Cannabidiol (CBD) cannabis oil as an adjunct therapy to methadone-based Opioid Agonist Therapy (OAT) for individuals with opioid use disorder (OUD) in a community setting.

DETAILED DESCRIPTION:
This is a single-site, two-phase pilot clinical trial evaluating the safety and feasibility of administering a balanced 1:1 ratio of THC:CBD cannabis oil alongside methadone-based opioid agonist therapy (OAT) in a community setting.

Phase 1 is a 12-week, double-blind, randomized controlled study involving 24 eligible participants with opioid use disorder (OUD) who recently initiated or re-initiated methadone-based OAT. Participants will be randomly assigned to receive either balanced THC:CBD cannabis oil or placebo oil. All participants will receive OUD clinical care, including OAT management, independent of research visits.

After the 12-week blinded treatment period (Phase 1), eligible participants will be invited to Phase 2, a 12-week open-label treatment extension study with all participants receiving balanced THC:CBD cannabis oil. Follow-up research visits will occur every two weeks from the start of open-label treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals of at least 25 years of age or older;
2. Diagnosed with OUD as per DSM-5 criteria;
3. Initiated or re-initiated methadone-based OAT within the past 30 days prior to study entry;
4. Cannabis-use experienced, defined as having used any amount of cannabis in the six months prior to the screening visit;
5. Willing to only use study-provided cannabis as directed by study protocol, including abstention from non-study cannabis and cannabinoids;
6. Agree to keep all study medication stored in a secure location and not to share/distribute study medication to any other individual;
7. If assigned female sex at birth:

   1. Be of non-childbearing potential, defined as (i) postmenopausal (12 months of spontaneous amenorrhea and over 45 years of age); or (ii) documented surgical sterilization (i.e., tubal ligation, hysterectomy, or bilateral oophorectomy); or
   2. If of childbearing potential, be willing to use an acceptable method of contraception throughout the study and have a negative pregnancy test at screening;
8. Ability to understand and comply with study protocol procedures and to provide written informed consent.

Inclusion criteria for Phase 2

In addition to meeting all eligibility criteria outlined in Phase 1, participants will be eligible for Phase 2 provided they meet ALL the following criteria at Week 12:

1. Participants who have not experienced a study medication-related serious adverse event during Phase 1;
2. Participants who have not been lost to follow-up during Phase 1.

Exclusion Criteria:

1. Any disabling, severe, or unstable medical or psychiatric condition that, in the opinion of the study physician, precludes safe participation in the study or the ability to provide fully informed consent, as assessed by medical and psychiatric history, physical examination, vital signs, and/or laboratory tests;
2. Any severe or unstable co-morbid substance use disorder (e.g., delirium tremens, acute alcohol intoxication) that, in the opinion of the study physician, precludes safe participation in the study;
3. Currently pregnant or breastfeeding, or planning to become pregnant;
4. Known or suspected allergy or hypersensitivity to cannabinoids;
5. History of respiratory disease, severe cardiovascular, cerebrovascular, renal or liver disease;
6. Current or historic cannabis use disorder;
7. Taking warfarin, clopidogrel, clobazam, theophylline, clozapine and olanzapine medications as they may interact with cannabinoids in a clinically significant manner if they cannot be switched to a different medication;
8. Any personal or family history (first degree relative) of primary psychotic disorders (i.e., schizophrenia, schizoaffective disorder) as per DSM-5 criteria;
9. Unable to abstain from driving any vehicle or operating machinery for at least 10 hours after taking the study medication. In cases where impairment persists beyond the initial 10-hour period, participants must continue to adhere to these restrictions until the impairment resolves;
10. Actively participating in other interventional clinical trial(s);
11. Incarcerated, pending legal action or other reasons that might prevent completion of the study.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 28 weeks
  The safety will be evaluated by monitoring and gathering information on physical exam, vital signs, pregnancy testing, adverse events (AE) and serious adverse events (SAE), from the screening visit up to the End of Treatment (EOT)/Early Termination visit. AEs and SAEs will be monitored and recorded throughout the study duration. The proportion of participants who experience AEs or SAEs will be assessed by study arm.
Risk of Treatment Contamination | 24 weeks
  The proportion of participants using non-study cannabis in the control arm, and proportion of days in Phase 1 where non-study cannabis was used. Self-report of non-study cannabis use will be collected using the Timeline Follow Back (TLFB).
Participants' adherence to treatment | 24 weeks
  The degree of compliance with the recommended treatment plan, including study drug dosage and administration. This measures how well participants are able to stick to the prescribed treatment regimen and whether or not they are able to complete the full course of treatment. This will be assessed through a self-reported measure, such as study drug diary or treatment logs.
Acceptability | 24 weeks
  Participant satisfaction with the assigned treatment will be assessed through administration of the Medical Safety Questionnaire (MSQ) every 4 weeks during treatment phase The MSQ is a participant-completed questionnaire that evaluates participant satisfaction with study treatment on a 7-point Likert scale.
Blinding effectiveness | 24 weeks
  The blinding success questionnaire will be used to evaluate the participants' awareness of their assigned treatment.
Adequacy of Dose | 24 weeks
  Patient satisfaction with dose level assessed through the adequacy of dose questionnaire and regular consultations

SECONDARY OUTCOMES:
The number of potential participants referred to the study | 24 weeks
The screening failure rates | 24 weeks
The monthly enrolment rates | 24 weeks
The proportion of eligible participants who are willing to be randomized, willing to initiate the intervention and willing to complete 12-week assessments by study arm | 24 weeks
The proportion of scheduled study visits completed by study arm | 24 weeks

OTHER OUTCOMES:
Retention in OAT | 24 weeks
  Retention in OAT will be measured by the proportion of participants on OAT at W12 and at W24, defined as having both a) an active OAT prescription at week 12/24, and b) a positive UDT result for the prescribed OAT at week 12/24.
Illicit opioid use | 24 weeks
  Suppression of illicit opioid use will be measured as the percentage of opioid-free weeks during W1-12, using a combination of Urine Drug Test (UDT) results and self-reported illicit opioid use assessed by the TLFB.
Pain Intensity | 24 weeks
  The severity of pain will be assessed by the validated scale within the Patient-Reported Outcomes Measurement Information System (PROMIS) 29+2 Profile v2.1 (PROPr): the PROMIS Pain Intensity item.
Pain Interference | 24 weeks
  The impact of pain on its impact on functioning will be assessed the validated scale within the Patient-Reported Outcomes Measurement Information System (PROMIS) 29+2 Profile v2.1 (PROPr): PROMIS SF v1.0 - Pain Interference 4a scale.
Anxiety | 24 weeks
  Anxiety symptoms will be assessed by the validated short scale within the PROMIS 29+2 Profile v2.1 (PROPr): the PROMIS SF v1.0 - Anxiety 4a
Depression | 24 weeks
  Depressive symptoms will be assessed by the validated short scale within the PROMIS 29+2 Profile v2.1 (PROPr): the PROMIS SF v1.0 - Depression 4a.
Changes in health-related quality of life | 24 weeks
  Changes in health-related quality of life (HRQoL) between screening and the end of treatment will be measured by the PROMIS 29+2 Profile v2.1 (PROPr).
Changes in substance-use related problems | 24 weeks
  The Addiction Severity Index (ASI) Self-Report form will be used to assess changes in substance-use related problems between Baseline (W0) prior to the start of treatment administration, Treatment Visit at W12 and EOT (W24)/Early Termination.
Opioid Craving | 24 weeks
  Opioid craving over time will be measured using a 100-mm visual analog scale (VAS), with 11 lines labeled from left to right with the numbers "0" to "10", and word anchors at each end representing the extremes, where "0=no craving" and "100 mm=most intense craving".

CONTACTS AND LOCATIONS:
Overall Officials: M Eugenia Socias, MD, MSc., Principal Investigator — Assistant Professor, Department of Medicine, University of British Columbia
Locations (1):
- Rapid Access Addiction Clinic (RAAC), St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No